CLINICAL TRIAL: NCT03588390
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Oral Doses of BI 1323495 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design)
Brief Title: This Study in Healthy Men Tests How Different Doses of BI 1323495 Are Taken up in the Body and How Well They Are Tolerated.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1405-0001; 2017-004899-62 (EudraCT Number)
Record Dates: First submitted 2018-07-06; First posted 2018-07-17 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Dose Group 1 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 1 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo
- Dose Group 2 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 2 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo
- Dose Group 3 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 3 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo
- Dose Group 4 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 4 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo
- Dose Group 5 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 5 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo
- Dose Group 6 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 6 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo
- Dose Group 7 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 7 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo
- Dose Group 8 (Experimental): Participants were orally administered single dose of BI 1323495 dose group 8 or matching placebo film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
  Interventions: Drug: BI 1323495; Drug: Placebo

INTERVENTIONS:
Drug: BI 1323495 — Low strength tablet
  Arms: Dose Group 1; Dose Group 2; Dose Group 3
Drug: BI 1323495 — Middle strength tablet
  Arms: Dose Group 4; Dose Group 5; Dose Group 6
Drug: BI 1323495 — High strength tablet
  Arms: Dose Group 7; Dose Group 8
Drug: Placebo — Placebo to low strength tablet
  Arms: Dose Group 1; Dose Group 2; Dose Group 3
Drug: Placebo — Placebo to middle strength tablet
  Arms: Dose Group 4; Dose Group 5; Dose Group 6
Drug: Placebo — Placebo to high strength tablet
  Arms: Dose Group 7; Dose Group 8

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1323495 in healthy male subjects following oral administration of single rising doses.

Secondary objectives are the exploration of the pharmacokinetics (PK) including dose proportionality and pharmacodynamics (PD) of BI 1323495 after single dosing and the assessment of the PK/PD relationship.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure [BP], Pulse Rate [PR]), 12-lead Electrocardiogram [ECG], and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index [BMI] of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice[ GCP] and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure [BP], Pulse Rate [PR] or Electrocardiogram [ECG]) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval such as QTc intervals that are repeatedly greater than 450 ms or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* Male subjects with female partner of childbearing potential who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication
* Current or history of relevant kidney, urinary tract diseases or abnormalities (e.g. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure)
* Estimated glomerular filtration rate according to CKD-EPI formula < 90 mL/min at screening
* Within 10 days prior to administration of trial medication, use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g., acetylsalicylic acid)
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. Studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement.

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-rising dose trial was designed as single-blind, partially randomised, and placebo-controlled within parallel dose groups.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist site which would then ensure that all participants met all strictly implemented inclusion/exclusion criteria. Participants were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- Placebo Matching BI 1323495: Participants were orally administered single dose of placebo matching to BI 1323495 film-coated tablets with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- BI 1323495 Dose Group 1: Participants were orally administered single dose of BI 1323495 dose group 1 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- BI 1323495 Dose Group 2: Participants were orally administered single dose of BI 1323495 dose group 2 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- BI 1323495 Dose Group 3: Participants were orally administered single dose of BI 1323495 dose group 3 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- BI 1323495 Dose Group 4: Participants were orally administered single dose of BI 1323495 dose group 4 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- BI 1323495 Dose Group 5: Participants were orally administered single dose of BI 1323495 dose group 5 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- BI 1323495 Dose Group 6: Participants were orally administered single dose of BI 1323495 dose group 6 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- BI 1323495 Dose Group 7: Participants were orally administered single dose of BI 1323495 dose group 7 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
- BI 1323495 Dose Group 8: Participants were orally administered single dose of BI 1323495 dose group 8 film-coated tablet with 240 mL of water after an overnight fast of at least 10 h.
Period: Overall Study
Arm/Group | Placebo Matching BI 1323495 | BI 1323495 Dose Group 1 | BI 1323495 Dose Group 2 | BI 1323495 Dose Group 3 | BI 1323495 Dose Group 4 | BI 1323495 Dose Group 5 | BI 1323495 Dose Group 6 | BI 1323495 Dose Group 7 | BI 1323495 Dose Group 8
Started | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who were documented to have received at least 1 dose of trial drug. It was used for analysis of safety, demographic data, and baseline characteristics, as well as for the description of biomarkers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 1323495 | BI 1323495 Dose Group 1 | BI 1323495 Dose Group 2 | BI 1323495 Dose Group 3 | BI 1323495 Dose Group 4 | BI 1323495 Dose Group 5 | BI 1323495 Dose Group 6 | BI 1323495 Dose Group 7 | BI 1323495 Dose Group 8 | Total
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.9 (6.0) | 28.0 (7.6) | 31.5 (6.4) | 29.8 (8.9) | 34.3 (5.4) | 33.7 (8.6) | 34.3 (6.5) | 30.8 (4.1) | 29.5 (5.2) | 30.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: Percentage of participants with drug-related adverse events.
Time Frame: From drug administration until end of trial, up to 15 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Matching BI 1323495 | BI 1323495 Dose Group 1 | BI 1323495 Dose Group 2 | BI 1323495 Dose Group 3 | BI 1323495 Dose Group 4 | BI 1323495 Dose Group 5 | BI 1323495 Dose Group 6 | BI 1323495 Dose Group 7 | BI 1323495 Dose Group 8
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of participants | 6.7 | 50.0 | 33.3 | 0.0 | 16.7 | 0.0 | 16.7 | 50.0 | 16.7

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 1323495 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) after single oral administration of BI 1323495.
Time Frame: 1 hour (h) before drug administration and 1, 2, 3, 4, 6, 7, 8, 9, 10, 12, 24, 34, 48, 72 and 96 h and additionally 4.75, 5.5, 6.5, 7.5 h for dose group 1/2/3 and 0.333, 0.667, 1.5, 5 h for dose group 4/5/6/7/8 after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This subject set included all subjects from the TS receiving BI 1323495 who provided at least 1 secondary PK parameter that was not excluded (due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)*hours (h) /Liter (L)
Arm/Group | BI 1323495 Dose Group 1 | BI 1323495 Dose Group 2 | BI 1323495 Dose Group 3 | BI 1323495 Dose Group 4 | BI 1323495 Dose Group 5 | BI 1323495 Dose Group 6 | BI 1323495 Dose Group 7 | BI 1323495 Dose Group 8
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanomole (nmol)*hours (h) /Liter (L) | 143 (102.0) | 883 (118.0) | 824 (77.7) | 2360 (73.5) | 3710 (69.4) | 3120 (140.0) | 1780 (102.0) | 3820 (71.9)
Statistical Analysis 1: Comparison: BI 1323495 Dose Group 1 vs BI 1323495 Dose Group 2 vs BI 1323495 Dose Group 3 vs BI 1323495 Dose Group 4 vs BI 1323495 Dose Group 5 vs BI 1323495 Dose Group 6 vs BI 1323495 Dose Group 7 vs BI 1323495 Dose Group 8; The basic model for the investigation of dose proportionality was a power model that described the functional relationship between the dose and PK endpoints; Test type: Other; Slope = 0.6960, 95% CI 2-sided [0.5006 to 0.8914], Standard Error of Mean 0.0971 — Based on the estimate for slope parameter (β), a 2-sided 95% CI for the slope was computed. Perfect dose proportionality would correspond to a slope of 1. Standard error of the mean is actually standard error of slope
Statistical Analysis 2: Comparison: BI 1323495 Dose Group 1 vs BI 1323495 Dose Group 2 vs BI 1323495 Dose Group 3 vs BI 1323495 Dose Group 4 vs BI 1323495 Dose Group 5 vs BI 1323495 Dose Group 6; [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 0.9244, 95% CI 2-sided [0.6764 to 1.1724], Standard Error of Mean 0.1220 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Maximum Measured Concentration of BI 1323495 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1323495 in plasma (Cmax) after single oral administration of BI 1323495.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 1323495 Dose Group 1 | BI 1323495 Dose Group 2 | BI 1323495 Dose Group 3 | BI 1323495 Dose Group 4 | BI 1323495 Dose Group 5 | BI 1323495 Dose Group 6 | BI 1323495 Dose Group 7 | BI 1323495 Dose Group 8
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol/L | 10.5 (66.3) | 59.4 (147.0) | 145.0 (74.8) | 229.0 (127.0) | 179.0 (152.0) | 136.0 (74.2) | 195.0 (90.8) | 195.0 (90.8)
Statistical Analysis 1: Comparison: BI 1323495 Dose Group 1 vs BI 1323495 Dose Group 2 vs BI 1323495 Dose Group 3 vs BI 1323495 Dose Group 4 vs BI 1323495 Dose Group 5 vs BI 1323495 Dose Group 6 vs BI 1323495 Dose Group 7 vs BI 1323495 Dose Group 8; [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 0.6533, 95% CI 2-sided [0.4556 to 0.8510], Standard Error of Mean 0.0982 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 1323495 Dose Group 1 vs BI 1323495 Dose Group 2 vs BI 1323495 Dose Group 3 vs BI 1323495 Dose Group 4 vs BI 1323495 Dose Group 5 vs BI 1323495 Dose Group 6; [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 0.8586, 95% CI 2-sided [0.5929 to 1.1242], Standard Error of Mean 0.1307 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From drug administration until end of trial, up to 15 days.
Description: Treated set (TS): This subject set included all subjects who were documented to have received at least 1 dose of trial drug. It was used for analysis of safety, demographic data, and baseline characteristics, as well as for the description of biomarkers.
Groups:
- Placebo Matching BI 1323495: Participants were orally administered single dose of placebo matching to BI 1323495 film-coated tablet with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- BI 1323495 Total: Participants were orally administered single dose of BI 1323495 dose groups 1, 2, 3, 4, 5, 6, 7 and 8 film-coated tablets with 240 mL of water after an overnight fast of at least 10 h.
Arm/Group | Placebo Matching BI 1323495 | BI 1323495 Dose Group 1 | BI 1323495 Dose Group 2 | BI 1323495 Dose Group 3 | BI 1323495 Dose Group 4 | BI 1323495 Dose Group 5 | BI 1323495 Dose Group 6 | BI 1323495 Dose Group 7 | BI 1323495 Dose Group 8 | BI 1323495 Total
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/48
Other Adverse Events (participants affected / at risk) | 2/15 | 3/6 | 2/6 | 1/6 | 2/6 | 1/6 | 2/6 | 3/6 | 2/6 | 16/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 1323495 (N=15) | BI 1323495 Dose Group 1 (N=6) | BI 1323495 Dose Group 2 (N=6) | BI 1323495 Dose Group 3 (N=6) | BI 1323495 Dose Group 4 (N=6) | BI 1323495 Dose Group 5 (N=6) | BI 1323495 Dose Group 6 (N=6) | BI 1323495 Dose Group 7 (N=6) | BI 1323495 Dose Group 8 (N=6) | BI 1323495 Total (N=48)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Unevaluable event (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Glutamate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT03588390/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03588390/SAP_001.pdf